CLINICAL TRIAL: NCT05069259
Title: A LOW-INTERVENTIONAL, PROSPECTIVE, MULTI-CENTER STUDY TO EVALUATE REAL-WORLD CLINICAL, BIOCHEMICAL AND PATIENT-REPORTED RESPONSES TO TOFACITINIB INDUCTION THERAPY IN PATIENTS WITH MODERATELY TO SEVERELY ACTIVE ULCERATIVE COLITIS IN SWITZERLAND
Brief Title: Generate Real World Data On Tofacitinib Induction Therapy and Changes In Clinical and Patient Reported Outcomes.
Acronym: KIC-START
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to difficulty in enrolling targeted number of participants. There were no safety and/or efficacy concerns in the decision to stop enrollment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921395; KIC-START (Other: Alias Study Number)
Record Dates: First submitted 2021-09-01; First posted 2021-10-06 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with active Ulcerative Colitis
  Interventions: Other: Stool sample collection

INTERVENTIONS:
Other: Stool sample collection — collection for measuring calprotectin levels

SUMMARY:
This study is expected to contribute to the body of real-world data of tofacitinib's safety and efficacy profile in ulcerative colitis. Conventional clinical outcomes will give a better understanding of response and remission rates in a representative, post-marketing population.

Regular patient questionnaires and measurement of a biomarker of gut inflammation will provide detail on how patients experience induction treatment and contextualise the efficacy data.

DETAILED DESCRIPTION:
This is a low-interventional study in which the intervention under study is home fecal calprotectin testing which falls outside of normal standard of care in ulcerative colitis. Tofacitinib is prescribed and administered as per the Swiss prescribing information. Accordingly, this study is registered on ClinicalTrials.gov as an interventional study. Under Swiss law, this study is considered and approved as a non-interventional study (Category A, Human Research Ordinance, Swiss Confederation).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years of age or older at screening visit
* Participants with confirmed diagnosis of UC and who are prescribed tofacitinib (Xeljanz®) for moderately to severely active UC as per the Swiss label
* Participants who are willing and able to comply with all scheduled visits, treatment plan, study interventions, and other study procedures
* Capable of giving personally signed informed consent

Exclusion Criteria:

* Presence of clinical findings suggestive of Crohn's disease
* Any previous exposure to tofacitinib including participation in the tofacitinib clinical program
* Co-medication with any other advanced therapies for UC (biologics*, azathioprine, mercaptopurine and methotrexate) or any other JAK inhibitor
* Any identified contra-indications for use of tofacitinib as per the Swiss label
* Not owning a handheld digital device compatible with the Sidekick Health App, not willing to have it installed on this device or not capable of using the App
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 adults both male and female who are prescribed tofacitinib for moderately to severely active UC will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Switzerland (5):
  - Kantonsspital St, Gallen, Sankt Gallen, Canton of St. Gallen
  - Clarunis, Universitätsspital, Basel
  - Verein IBD Study Group, Bern
  - Centre Fribourgeois de Gastroenterologie, Fribourg
  - Kantonsspital Baselland, Liestal

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderately to severely active ulcerative colitis (UC) who were prescribed tofacitinib in real world setting as routine clinical practice across Switzerland were enrolled in this study.
Groups:
- All Participants: Participants with moderately to severely active UC who were prescribed tofacitinib by the treating physician in routine clinical practice as per the Swiss prescribing information, were included.
Period: Overall Study
Arm/Group | All Participants
Started | 18
Completed | 16
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Sponsor decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 41 [30 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Response at Week 8
Description: Clinical response was defined as a reduction in the partial Mayo score (PMS) from baseline of >=2 points or achieving clinical remission. Clinical remission was defined as PMS of <= 2 with no subscore >1. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity.
Time Frame: Week 8
Population: Full analysis set (FAS) included all participants who were included in the study (i.e., performed baseline visit and received a study identification number). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 16
Percentage of participants | 63 [39 to 82]

2. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 8
Description: Clinical remission was defined as PMS of <= 2 with no subscore >1. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity.
Time Frame: Week 8
Population: FAS included all participants who were included in the study (i.e., performed baseline visit and received a study identification number). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 16
Percentage of participants | 38 [18 to 61]

3. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response at Week 16
Description: Clinical response was defined as a reduction in the PMS from baseline of >=2 points or achieving clinical remission. Clinical remission was defined as PMS of <= 2 with no subscore >1. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
Percentage of participants | 73 [48 to 89]

4. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
Percentage of participants | 40 [20 to 64]

5. Secondary Outcome: Percentage of Participants Who Achieved Inflammatory Bowel Disease Questionnaire (IBDQ) Remission at Week 8
Description: IBDQ remission was defined as an IBDQ score >= 170. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 13
Percentage of participants | 46 [23 to 71]

6. Secondary Outcome: Percentage of Participants Who Achieved IBDQ Remission at Week 16
Description: as for outcome 5
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 7
Percentage of participants | 71 [36 to 92]

7. Secondary Outcome: Percentage of Participants Who Achieved IBDQ Response at Week 8
Description: IBDQ response was defined as an IBDQ score >=16 points higher than IBDQ baseline score. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 13
Percentage of participants | 69 [42 to 87]

8. Secondary Outcome: Percentage of Participants Who Achieved IBDQ Response at Week 16
Description: as for outcome 7
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 7
Percentage of participants | 100 [65 to 100]

9. Secondary Outcome: Percentage of Participants Who Achieved Biochemical Remission at Week 8
Description: Biochemical remission was defined as a fecal calprotectin (fCAL) concentration <=250 micrograms per gram (mcg/g). fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 9
Percentage of participants | 11 [2.0 to 43]

10. Secondary Outcome: Percentage of Participants Who Achieved Biochemical Remission at Week 16
Description: Biochemical remission was defined as a fCAL concentration <=250 mcg/g. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 6
Percentage of participants | 33 [9.7 to 70]

11. Secondary Outcome: Median Change From Baseline in Stool Frequency Measured by Mayo Score Stool Frequency Subscore at Weeks 8 and 16
Description: The stool frequency patient reported outcome (PRO) was assessed with one question about the number of stools on a given day. The Mayo Score stool frequency subscore was used for scoring. Scores ranged from 0 to 3 (0= normal number of stools; 1= 1-2 stools more than normal; 2= 3-4 stools more than normal and 3= 5 or more stools than normal) where higher scores indicated more severe disease activity.
Time Frame: Baseline, Week 8 and Week 16
Population: FAS included all participants who were included in the study (i.e., performed baseline visit and received a study identification number). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for specified rows. All participants under "Overall Number of Participants Analyzed" contributed data to the table but may not have data evaluable for every row.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score on a scale
  Change at Week 8: number analyzed (Participants) | 13
  Change at Week 8 | 0 [-1 to 1]
  Change at Week 16: number analyzed (Participants) | 7
  Change at Week 16 | -1 [-2 to -1]

12. Secondary Outcome: Median Change From Baseline in Rectal Bleeding Measured by Mayo Score Rectal Bleeding Subscore at Weeks 8 and 16
Description: The rectal bleeding PRO was assessed with one question about most severe rectal bleeding on a given day. The Mayo Score rectal bleeding subscore was used for scoring. Scores ranged from 0 to 3 (0= no blood seen; 1= streaks of blood with stool less than half the time; 2= obvious blood with stool most of the time and 3= blood alone passes) where higher scores indicated more severe bleeding of the day.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score on a scale
  Change at Week 8: number analyzed (Participants) | 13
  Change at Week 8 | 0 [0 to 0]
  Change at Week 16: number analyzed (Participants) | 7
  Change at Week 16 | 0 [-1 to 0]

13. Secondary Outcome: Median Change From Baseline in Urgency of Defecation Assessed Using Numeric Rating Scale (NRS) at Weeks 8 and 16
Description: The urgency of defecation was assessed with the urgency NRS. Scoring was done on a 11-point NRS. Participant provided a score from 0 (no urgency) to 10 (worst possible urgency). Higher scores indicated more severe urgency.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score on a scale
  Change at Week 8: number analyzed (Participants) | 13
  Change at Week 8 | -1 [-2 to 0]
  Change at Week 16: number analyzed (Participants) | 7
  Change at Week 16 | -2 [-4 to -2]

14. Secondary Outcome: Median Change From Baseline in Abdominal Pain Assessed Using Pain NRS at Weeks 8 and 16
Description: The abdominal pain was assessed with the pain NRS. Scoring was done on a 10-point horizontal NRS. Participant provided a score from 1 (none) to 10 (very severe). Higher scores indicated more severe pain.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score on a scale
  Change at Week 8: number analyzed (Participants) | 14
  Change at Week 8 | -1 [-2 to 0]
  Change at Week 16: number analyzed (Participants) | 7
  Change at Week 16 | -2 [-3 to -1]

15. Secondary Outcome: Median Change From Baseline in Quality of Sleep Assessed Using NRS at Weeks 8 and 16
Description: The quality of sleep was assessed with a question from the sleep quality visual analogue scale survey. Scoring was done on a 11 NRS. Participant provided a score from 0 (very bad) to 10 (great). Higher scores indicated better quality of sleep.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score on a scale
  Change at Week 8: number analyzed (Participants) | 13
  Change at Week 8 | 2 [0 to 3]
  Change at Week 16: number analyzed (Participants) | 8
  Change at Week 16 | 3 [0 to 3]

16. Secondary Outcome: Median Change From Baseline in Daily Fatigue Assessed Using NRS at Weeks 8 and 16
Description: The daily fatigue was assessed with the fatigue NRS. Scoring was done on a 11-point NRS. Participant provided a score from 0 (no fatigue) to 10 (as bad as you can imagine). Higher scores indicated more severe fatigue.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score on a scale
  Change at Week 8: number analyzed (Participants) | 13
  Change at Week 8 | -1 [-3 to -1]
  Change at Week 16: number analyzed (Participants) | 8
  Change at Week 16 | -3 [-4 to -1]

17. Secondary Outcome: Median Change From Baseline in Weekly Fatigue Assessed Using FACIT-F at Weeks 8 and 16
Description: The weekly fatigue was assessed with 13 questions from the functional assessment of chronic illness therapy - fatigue (FACIT-F) version (v)4. Participants rated the intensity of their fatigue symptoms on a scale of 0 (not at all) to 4 (very much) for each 13 questions. Total score ranged from 0 to 52, with higher scores representing lower fatigue.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score on a scale
  Change at Week 8: number analyzed (Participants) | 13
  Change at Week 8 | 12 [-1 to 14]
  Change at Week 16: number analyzed (Participants) | 7
  Change at Week 16 | 13 [11 to 20]

18. Secondary Outcome: Median Change From Baseline in IBDQ Score (Total) at Weeks 8 and 16
Description: The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score on a scale
  Change at Week 8: number analyzed (Participants) | 13
  Change at Week 8 | 35 [11 to 54]
  Change at Week 16: number analyzed (Participants) | 7
  Change at Week 16 | 48 [44 to 77]

19. Secondary Outcome: Median Change From Baseline in fCAL at Weeks 8 and 16
Description: fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: micrograms per gram
Arm/Group | All Participants
Number analyzed (Participants) | 15
micrograms per gram
  Change at Week 8: number analyzed (Participants) | 9
  Change at Week 8 | -44 [-392 to -12]
  Change at Week 16: number analyzed (Participants) | 6
  Change at Week 16 | -24 [-78 to 267]

20. Secondary Outcome: Correlations Between PMS and IBDQ Score
Description: Correlation between PMS and IBDQ score was assessed by Spearman correlation coefficient. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Baseline, Week 8 and Week 16
Population: FAS included all participants who were included in the study (i.e., performed baseline visit and received a study identification number). Here, "Number Analyzed" signifies participants evaluable for specified rows. All participants under "Overall Number of Participants Analyzed" contributed data to the table but may not have data evaluable for every row.
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 16
  Baseline | -0.5
  Week 8: number analyzed (Participants) | 13
  Week 8 | -0.8
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.5

21. Secondary Outcome: Correlations Between PMS and fCAL Concentration
Description: Correlation between PMS and fCAL concentration was assessed by Spearman correlation coefficient. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0.4
  Week 8: number analyzed (Participants) | 9
  Week 8 | 0.1
  Week 16: number analyzed (Participants) | 6
  Week 16 | -0.8

22. Secondary Outcome: Correlations Between Stool Frequency and fCAL Concentration
Description: Correlation between stool frequency PRO and fCAL concentration was assessed by Spearman correlation coefficient. The stool frequency PRO was assessed with one question about the number of stools on a given day. The mayo score stool frequency subscore was used for scoring. Scores ranged from 0 to 3 (0= normal number of stools; 1= 1-2 stools more than normal; 2= 3-4 stools more than normal and 3= 5 or more stools than normal) where higher scores indicated more severe disease activity. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0.5
  Week 8: number analyzed (Participants) | 9
  Week 8 | 0
  Week 16: number analyzed (Participants) | 6
  Week 16 | -0.3

23. Secondary Outcome: Correlations Between Rectal Bleeding and fCAL Concentration
Description: Correlation between rectal bleeding PRO and fCAL concentration was assessed by Spearman correlation coefficient. The rectal bleeding PRO was assessed with one question about most severe rectal bleeding on a given day. The Mayo Score rectal bleeding subscore was used for scoring. Scores ranged from 0 to 3 (0= no blood seen; 1= streaks of blood with stool less than half the time; 2= obvious blood with stool most of the time and 3= blood alone passes) where higher scores indicated more severe bleeding of the day. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0.2
  Week 8: number analyzed (Participants) | 9
  Week 8 | 0.4
  Week 16: number analyzed (Participants) | 5
  Week 16 | -0.4

24. Secondary Outcome: Correlations Between Urgency of Defecation and fCAL Concentration
Description: Correlation between urgency of defecation and fCAL concentration was assessed by Spearman correlation coefficient. The urgency of defecation was assessed with the urgency NRS. Scoring was done on a 11-point NRS. Participant provided a score from 0 (no urgency) to 10 (worst possible urgency). Higher scores indicated more severe urgency. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0.2
  Week 8: number analyzed (Participants) | 9
  Week 8 | 0.1
  Week 16: number analyzed (Participants) | 5
  Week 16 | -0.2

25. Secondary Outcome: Correlations Between Abdominal Pain and fCAL Concentration
Description: Correlation between abdominal pain and fCAL was assessed by Spearman correlation coefficient. The abdominal pain was assessed with the pain NRS. Scoring was done on a 10-point horizontal NRS. Participant provided a score from 1 (none) to 10 (very severe). Higher scores indicated more severe pain. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0.4
  Week 8: number analyzed (Participants) | 9
  Week 8 | 0
  Week 16: number analyzed (Participants) | 5
  Week 16 | 0.3

26. Secondary Outcome: Correlations Between Quality of Sleep and fCAL Concentration
Description: Correlation between quality of sleep and fCAL concentration was assessed by Spearman correlation coefficient. The quality of sleep was assessed with a question from the sleep quality visual analogue scale survey. Scoring was done on a 11-point NRS. Participant provided a score from 0 (very bad) to 10 (great). Higher scores indicated better quality of sleep. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0
  Week 8: number analyzed (Participants) | 9
  Week 8 | -0.2
  Week 16: number analyzed (Participants) | 5
  Week 16 | 0

27. Secondary Outcome: Correlations Between Daily Fatigue and fCAL Concentration
Description: Correlation between daily fatigue and fCAL concentration was assessed by Spearman correlation coefficient. The daily fatigue was assessed with the fatigue NRS. Scoring was done on a 11-point NRS. Participant provided a score from 0 (no fatigue) to 10 (as bad as you can imagine). Higher scores indicated more severe fatigue. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | -0.1
  Week 8: number analyzed (Participants) | 9
  Week 8 | -0.1
  Week 16: number analyzed (Participants) | 5
  Week 16 | 0.2

28. Secondary Outcome: Correlations Between Weekly Fatigue and fCAL Concentration
Description: Correlation between weekly fatigue and fCAL concentration was assessed by Spearman correlation coefficient. The weekly fatigue was assessed with 13 questions from the FACIT-F v4. Participants rated the intensity of their fatigue symptoms on a scale of 0 (not at all) to 4 (very much) for each 13 questions. Total score ranged from 0 to 52, with higher scores representing lower fatigue. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 14
  Baseline | 0.2
  Week 8: number analyzed (Participants) | 9
  Week 8 | 0.5
  Week 16: number analyzed (Participants) | 5
  Week 16 | -0.9

29. Secondary Outcome: Correlations Between IBDQ Score and fCAL Concentration
Description: Correlation between IBDQ score and fCAL concentration was assessed by Spearman correlation coefficient. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life. fCAL is a small anti-microbial protein detected in stool that constitutes approximately 60% of neutrophil cytoplasm. As migration of neutrophils into the intestinal mucosa is a hallmark of active intestinal inflammation, fCAL serves as a non-invasive biomarker for intestinal inflammation.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | -0.4
  Week 8: number analyzed (Participants) | 9
  Week 8 | -0.1
  Week 16: number analyzed (Participants) | 5
  Week 16 | 0.2

30. Secondary Outcome: Correlations Between Stool Frequency and IBDQ Score
Description: Correlation between stool frequency PRO and IBDQ score was assessed by Spearman correlation coefficient. The stool frequency PRO was assessed with one question about the number of stools on a given day. The Mayo Score stool frequency subscore was used for scoring. Scores ranged from 0 to 3 (0= normal number of stools; 1= 1-2 stools more than normal; 2= 3-4 stools more than normal and 3= 5 or more stools than normal) where higher scores indicated more severe disease activity. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | -0.3
  Week 8: number analyzed (Participants) | 13
  Week 8 | -0.7
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.3

31. Secondary Outcome: Correlations Between Rectal Bleeding and IBDQ Score
Description: Correlation between rectal bleeding PRO and IBDQ score was assessed by Spearman correlation coefficient. The rectal bleeding PRO was assessed with one question about most severe rectal bleeding on a given day. The Mayo Score rectal bleeding subscore was used for scoring. Scores ranged from 0 to 3 (0= no blood seen; 1= streaks of blood with stool less than half the time; 2= obvious blood with stool most of the time and 3= blood alone passes) where higher scores indicated more severe bleeding of the day. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | -0.5
  Week 8: number analyzed (Participants) | 13
  Week 8 | -0.6
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.6

32. Secondary Outcome: Correlations Between Urgency of Defecation and IBDQ Score
Description: Correlation between urgency of defecation and IBDQ score was assessed by Spearman correlation coefficient. The urgency of defecation was assessed with the urgency NRS. Scoring was done on a 11-point NRS. Participant provided a score from 0 (no urgency) to 10 (worst possible urgency). Higher scores indicated more severe urgency. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | -0.7
  Week 8: number analyzed (Participants) | 13
  Week 8 | -0.9
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.1

33. Secondary Outcome: Correlations Between Abdominal Pain and IBDQ Score
Description: Correlation between abdominal pain and IBDQ score was assessed by Spearman correlation coefficient. The abdominal pain was assessed with the pain NRS. Scoring was done on a 10-point horizontal NRS. Participant provided a score from 1 (none) to 10 (very severe). Higher scores indicated more severe pain. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 16
  Baseline | -0.6
  Week 8: number analyzed (Participants) | 13
  Week 8 | -0.9
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.5

34. Secondary Outcome: Correlations Between Quality of Sleep and IBDQ Score
Description: Correlation between quality of sleep and IBDQ score was assessed by Spearman correlation coefficient. The quality of sleep was assessed with a question from the sleep quality visual analogue scale survey. Scoring was done on a 11-point NRS. Participant provided a score from 0 (very bad) to 10 (great). Higher scores indicated better quality of sleep. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 16
  Baseline | 0.3
  Week 8: number analyzed (Participants) | 13
  Week 8 | 0.5
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.4

35. Secondary Outcome: Correlations Between Daily Fatigue and IBDQ Score
Description: Correlation between daily fatigue and IBDQ score was assessed by Spearman correlation coefficient. The daily fatigue was assessed with the fatigue NRS. Scoring was done on a 11-point NRS. Participant provided a score from 0 (no fatigue) to 10 (as bad as you can imagine). Higher scores indicated more severe fatigue. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0
  Week 8: number analyzed (Participants) | 13
  Week 8 | -0.8
  Week 16: number analyzed (Participants) | 7
  Week 16 | 0.2

36. Secondary Outcome: Correlations Between Weekly Fatigue and IBDQ Score
Description: Correlation between weekly fatigue and IBDQ score was assessed by Spearman correlation coefficient. The weekly fatigue was assessed with 13 questions from the FACIT-F v4. Participants rated the intensity of their fatigue symptoms on a scale of 0 (not at all) to 4 (very much) for each 13 questions. Total score ranged from 0 to 52, with higher scores representing lower fatigue. The IBDQ was a 32-item questionnaire grouped into four dimensions: bowel symptoms, systemic symptoms, emotional function and social function, where range was as follows: bowel symptoms: 10 to 70; systemic symptoms: 5 to 35; emotional function: 12 to 84 and social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicated better quality of life.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 16
  Baseline | 0.3
  Week 8: number analyzed (Participants) | 13
  Week 8 | 0.7
  Week 16: number analyzed (Participants) | 7
  Week 16 | 0.1

37. Secondary Outcome: Correlations Between PMS and Stool Frequency
Description: Correlation between PMS and stool frequency PRO was assessed by Spearman correlation coefficient. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. The stool frequency PRO was assessed with one question about the number of stools on a given day. The Mayo Score stool frequency subscore was used for scoring. Scores ranged from 0 to 3 (0= normal number of stools; 1= 1-2 stools more than normal; 2= 3-4 stools more than normal and 3= 5 or more stools than normal) where higher scores indicated more severe disease activity.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0.6
  Week 8: number analyzed (Participants) | 13
  Week 8 | 0.8
  Week 16: number analyzed (Participants) | 7
  Week 16 | 0.4

38. Secondary Outcome: Correlations Between PMS and Rectal Bleeding
Description: Correlation between PMS and rectal bleeding PRO was assessed by Spearman correlation coefficient. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. The rectal bleeding PRO was assessed with one question about most severe rectal bleeding on a given day. The Mayo Score rectal bleeding subscore was used for scoring. Scores ranged from 0 to 3 (0= no blood seen; 1= streaks of blood with stool less than half the time; 2= obvious blood with stool most of the time and 3= blood alone passes) where higher scores indicated more severe bleeding of the day.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0.6
  Week 8: number analyzed (Participants) | 13
  Week 8 | 0.6
  Week 16: number analyzed (Participants) | 7
  Week 16 | 0.7

39. Secondary Outcome: Correlations Between PMS and Urgency of Defecation
Description: Correlation between PMS and urgency of defecation was assessed by Spearman correlation coefficient. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. The urgency of defecation was assessed with the urgency NRS. Scoring was done on a 11-point NRS. Participant provided a score from 0 (no urgency) to 10 (worst possible urgency). Higher scores indicated more severe urgency.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | 0.4
  Week 8: number analyzed (Participants) | 13
  Week 8 | 0.7
  Week 16: number analyzed (Participants) | 7
  Week 16 | 0.1

40. Secondary Outcome: Correlations Between PMS and Abdominal Pain
Description: Correlation between PMS and abdominal pain was assessed by Spearman correlation coefficient. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. The abdominal pain was assessed with the pain NRS. Scoring was done on a 10-point horizontal NRS. Participant provided a score from 1 (none) to 10 (very severe). Higher scores indicated more severe pain.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 16
  Baseline | 0.4
  Week 8: number analyzed (Participants) | 14
  Week 8 | 0.6
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.1

41. Secondary Outcome: Correlations Between PMS and Quality of Sleep
Description: Correlation between PMS and quality of sleep was assessed by Spearman correlation coefficient. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. The quality of sleep was assessed with a question from the sleep quality visual analogue scale survey. Scoring was done on a 11-point NRS. Participant provided a score from 0 (very bad) to 10 (great). Higher scores indicated better quality of sleep.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 16
  Baseline | -0.1
  Week 8: number analyzed (Participants) | 13
  Week 8 | -0.5
  Week 16: number analyzed (Participants) | 8
  Week 16 | 0.4

42. Secondary Outcome: Correlations Between PMS and Daily Fatigue
Description: Correlation between PMS and daily fatigue was assessed by Spearman correlation coefficient. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. The daily fatigue was assessed with the fatigue NRS. Scoring was done on a 11-point NRS. Participant provided a score from 0 (no fatigue) to 10 (as bad as you can imagine). Higher scores indicated more severe fatigue.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 15
  Baseline | -0.1
  Week 8: number analyzed (Participants) | 13
  Week 8 | 0.6
  Week 16: number analyzed (Participants) | 8
  Week 16 | -0.4

43. Secondary Outcome: Correlations Between PMS and Weekly Fatigue
Description: Correlation between PMS and weekly fatigue was assessed by Spearman correlation coefficient. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. The weekly fatigue was assessed with 13 questions from the FACIT-F v4. Participants rated the intensity of their fatigue symptoms on a scale of 0 (not at all) to 4 (very much) for each 13 questions. Total score ranged from 0 to 52, with higher scores representing lower fatigue.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 20
Measure: Number; unit: Correlation Coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 18
Correlation Coefficient
  Baseline: number analyzed (Participants) | 16
  Baseline | -0.2
  Week 8: number analyzed (Participants) | 13
  Week 8 | -0.6
  Week 16: number analyzed (Participants) | 7
  Week 16 | 0.6

44. Secondary Outcome: Median fCAL Concentrations Over Time Stratified by Week 8 Clinical Remission Status
Description: Clinical remission was defined as PMS of <= 2 with no subscore >1. Partial mayo score consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. In this outcome measure, fCAL concentration are reported at specified time points in those participants who had clinical remission at Week 8 and in those participants who did not have clinical remission at Week 8.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: micrograms per gram
Arm/Group | All Participants
Number analyzed (Participants) | 16
micrograms per gram
  fCAL concentrations at baseline in participants with clinical remission at Week 8: number analyzed (Participants) | 6
  fCAL concentrations at baseline in participants with clinical remission at Week 8 | 590 [297 to 616]
  fCAL concentrations at week 8 in participants with clinical remission at Week 8: number analyzed (Participants) | 4
  fCAL concentrations at week 8 in participants with clinical remission at Week 8 | 466 [253 to 638]
  fCAL concentrations at week 16 in participants with clinical remission at Week 8: number analyzed (Participants) | 2
  fCAL concentrations at week 16 in participants with clinical remission at Week 8 | 788 [681 to 894]
  fCAL concentrations at baseline in participants without clinical remission at Week 8: number analyzed (Participants) | 8
  fCAL concentrations at baseline in participants without clinical remission at Week 8 | 622 [376 to 984]
  fCAL concentrations at week 8 in participants without clinical remission at Week 8: number analyzed (Participants) | 5
  fCAL concentrations at week 8 in participants without clinical remission at Week 8 | 586 [581 to 593]
  fCAL concentrations at week 16 in participants without clinical remission at Week 16: number analyzed (Participants) | 4
  fCAL concentrations at week 16 in participants without clinical remission at Week 16 | 201 [64 to 498]

45. Secondary Outcome: Median fCAL Concentrations Over Time Stratified by Week 16 Clinical Remission Status
Description: Clinical remission was defined as PMS of <= 2 with no subscore >1. Partial mayo score consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. In this outcome measure, fCAL concentration are reported at specified time points in those participants who had clinical remission at Week 16 and in those participants who did not have clinical remission at Week 16.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: micrograms per gram
Arm/Group | All Participants
Number analyzed (Participants) | 15
micrograms per gram
  fCAL concentrations at baseline in participants with clinical remission at Week 16: number analyzed (Participants) | 6
  fCAL concentrations at baseline in participants with clinical remission at Week 16 | 612 [304 to 633]
  fCAL concentrations at week 8 in participants with clinical remission at Week 16: number analyzed (Participants) | 5
  fCAL concentrations at week 8 in participants with clinical remission at Week 16 | 586 [324 to 593]
  fCAL concentrations at week 16 in participants with clinical remission at Week 16: number analyzed (Participants) | 3
  fCAL concentrations at week 16 in participants with clinical remission at Week 16 | 1000 [788 to 1000]
  fCAL concentrations at baseline in participants without clinical remission at Week 16: number analyzed (Participants) | 7
  fCAL concentrations at baseline in participants without clinical remission at Week 16 | 607 [328 to 903]
  fCAL concentrations at week 8 in participants without clinical remission at Week 16: number analyzed (Participants) | 4
  fCAL concentrations at week 8 in participants without clinical remission at Week 16 | 642 [581 to 708]
  fCAL concentrations at week 16 in participants without clinical remission at Week 16: number analyzed (Participants) | 3
  fCAL concentrations at week 16 in participants without clinical remission at Week 16 | 71 [58 to 201]

46. Secondary Outcome: Median fCAL Concentrations Over Time Stratified by Week 8 Clinical Response Status
Description: Clinical response was defined as a reduction in the PMS from baseline of >=2 points or achieving clinical remission. Clinical remission was defined as PMS of <= 2 with no subscore >1. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. In this outcome measure, fCAL concentration are reported at specified time points in those participants who had clinical response at Week 8 and in those participants who did not have clinical response at Week 8.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: micrograms per gram
Arm/Group | All Participants
Number analyzed (Participants) | 16
micrograms per gram
  fCAL concentrations at baseline in participants with clinical response at Week 8: number analyzed (Participants) | 10
  fCAL concentrations at baseline in participants with clinical response at Week 8 | 501 [211 to 616]
  fCAL concentrations at week 8 in participants with clinical response at Week 8: number analyzed (Participants) | 6
  fCAL concentrations at week 8 in participants with clinical response at Week 8 | 597 [390 to 679]
  fCAL concentrations at week 16 in participants with clinical response at Week 8: number analyzed (Participants) | 5
  fCAL concentrations at week 16 in participants with clinical response at Week 8 | 331 [71 to 575]
  fCAL concentrations at baseline in participants without clinical response at Week 8: number analyzed (Participants) | 4
  fCAL concentrations at baseline in participants without clinical response at Week 8 | 819 [630 to 1000]
  fCAL concentrations at week 8 in participants without clinical response at Week 8: number analyzed (Participants) | 3
  fCAL concentrations at week 8 in participants without clinical response at Week 8 | 581 [581 to 587]
  fCAL concentrations at week 16 in participants without clinical response at Week 8: number analyzed (Participants) | 1
  fCAL concentrations at week 16 in participants without clinical response at Week 8 | 1000 [1000 to 1000]

47. Secondary Outcome: Median fCAL Concentrations Over Time Stratified by Week 16 Clinical Response Status
Description: Clinical response was defined as a reduction in the PMS from baseline of >=2 points or achieving clinical remission. Clinical remission was defined as PMS of <= 2 with no subscore >1. PMS consisted of 3 components: rectal bleeding, stool frequency, and physician global assessment of disease activity. Each sub score ranged from 0 (normal) to 3 (extreme severity). These sub scores were summed up to give a total score range of 0 (normal) to 9 (extreme severity), where higher scores indicated more disease severity. In this outcome measure, fCAL concentration are reported at specified time points in those participants who had clinical response at Week 16 and in those participants who did not have clinical response at Week 16.
Time Frame: Baseline, Week 8 and Week 16
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: micrograms per gram
Arm/Group | All Participants
Number analyzed (Participants) | 15
micrograms per gram
  fCAL concentrations at baseline in participants with clinical response at Week 16: number analyzed (Participants) | 9
  fCAL concentrations at baseline in participants with clinical response at Week 16 | 603 [204 to 637]
  fCAL concentrations at week 8 in participants with clinical response at Week 16: number analyzed (Participants) | 5
  fCAL concentrations at week 8 in participants with clinical response at Week 16 | 586 [324 to 593]
  fCAL concentrations at week 16 in participants with clinical response at Week 16: number analyzed (Participants) | 5
  fCAL concentrations at week 16 in participants with clinical response at Week 16 | 575 [71 to 1000]
  fCAL concentrations at baseline in participants without clinical response at Week 16: number analyzed (Participants) | 4
  fCAL concentrations at baseline in participants without clinical response at Week 16 | 706 [562 to 854]
  fCAL concentrations at week 8 in participants without clinical response at Week 16: number analyzed (Participants) | 4
  fCAL concentrations at week 8 in participants without clinical response at Week 16 | 642 [581 to 708]
  fCAL concentrations at week 16 in participants without clinical response at Week 16: number analyzed (Participants) | 1
  fCAL concentrations at week 16 in participants without clinical response at Week 16 | 331 [331 to 331]

ADVERSE EVENTS:
Time Frame: Maximum up to 20 weeks
Description: Same event may appear as both AE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. FAS included all participants who were included in the study (i.e., performed baseline visit and received a study identification number).
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 4/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=18)
Worsening Ulcerative Colitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=18)
Worsening Ulcerative Colitis (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Shingles (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT05069259/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT05069259/SAP_001.pdf